CLINICAL TRIAL: NCT04536831
Title: The Association of Vitamin D Supplementation With the Outcome in Critically Ill Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Mustahsin Khalil (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Sponsor-Investigator, Dr Mustahsin Khalil, Post graduate Trainee, King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: MKA1
Record Dates: First submitted 2020-08-21; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Critically Ill
Keywords: vitamin D; Supplimentation; Critically ill children
MeSH Terms: conditions — Critical Illness | interventions — Vitamin D; Cholecalciferol; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental): Consisted of 48 patients selected on admission via lottery method those will be given Vitamin D mega dose
  Interventions: Drug: Vitamin D
- Normal Saline group (Placebo Comparator): Consisted of 48 patients selected on admission via lottery method those will be given Normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Vitamin D — Vitamin D will be given to group A selected by Lottery method
  Other Names: vitamin D3
  Arms: Vitamin D group
Drug: Normal saline — Vitamin D will be given to group B slected by Lottery method
  Arms: Normal Saline group

SUMMARY:
Vitamin D deficiency is highly prevalent in critically ill adult and pediatric population that causes multiple adverse health outcomes including higher illness severity score, increased morbidity and mortality, multiple organ dysfunction, longer duration of Mechanical ventilation, longer duration of Oxygen therapy and increased length of stay (LOS) in PICU and hospital. Vitamin D deficiency is a modifiable risk factor that can be corrected with high dose of vitamin D supplementation to improve the clinical outcome.

This study is designed to determine whether random vitamin D supplementation within dose limits improves clinical outcomes in critically ill children.

DETAILED DESCRIPTION:
Vitamin D is known for its role in bone metabolism and calcium haemostasis but it is also required for the optimal functioning of cardiovascular and innate immune systems.

As a pleiotropic hormone it has been increasingly implicated in proper functioning of multiple organs; its deficiency is associated with cardiovascular diseases, asthma, cancer, multiple sclerosis, diabetes and acute lower respiratory tract infections. Over one billion people are vitamin D deficient worldwide and in Pakistani population vitamin D deficiency is reported as high as 76% despite abundant sunshine.

Beside of ambulatory individuals, the patients presenting in intensive care units are also found Vitamin D deficient. In adult intensive care settings studies have shown vitamin D deficiency (VDD) present in 60% of critically ill adult patients.VDD is also very common in pediatric intensive care units (PICU) worldwide, ranging from 30 to 80%.

Although there is high prevalence of VDD in pediatric and adult population, but there is no uniform definition of VDD exists. Levels of active metabolite 1,25(OH)2D of Vitamin D at tissue level cannot be measured, however, patient's blood level of 25-hydroxy vitamin D is used to know vitamin D stores in the body. Patient with serum vitamin D level<20ng/ml is considered to be vitamin D deficient.

VDD is associated with clinically poor outcomes like increased duration of mechanical ventilation, increased length of hospital stay, Sepsis, Acute respiratory failure and mortality in critically ill patients.

The existing evidences suggest that Vitamin D3 supplementation enhances recovery from influenza, recurrent pneumonias and tuberculosis. Recently, an observational study of adult patients suggested that patients with VDD showed decrease in the odds of all cause-mortality when their Vitamin D status was improved before hospitalization.

A randomized study demonstrated that one time bolus dose of oral vitamin D supplementation caused decrease in mortality in a group of patients with severe VDD.

A significant literature is available that suggests vitamin D deficiency as a modifiable risk factor in PICU settings. The recognized importance of vitamin D to the health of multiple organ systems suggest that rapid normalization could represent a simple, inexpensive, and safe means of improving outcomes and reducing health care spending.

This study is designed to supplement large dose of vitamin D that may lead to fast correction of low vitamin D level in critically ill children and possibility of better clinical outcome. If such an association is established by this study, routine detection and use of Vitamin D might be recommended for critically ill children admitted to PICU.

ELIGIBILITY:
Inclusion Criteria:

• Children of age 6 months to 10 years, either gender admitted in ICU for critical illness (on medical record) with PIM-2 score suggesting probability of mortality more than 50%.

Exclusion Criteria:

* Children with known adrenal, pituitary, hypothalamic or thyroid disease.
* Those who have complex congenital defects.
* Moribund at time of admission.
* Those who were expected to be care withdrawn.
* Patients who had received large dose regimen (200,000 IU or more) of vitamin D during the previous three months before admission.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Death | upto one month
  Patient is declared dead by duty doctor
Discharge | upto one month
  Patient became vitally stable and shifted out of PICU

SECONDARY OUTCOMES:
Duration of O2 therapy | upto one month
  Total time that patient required O2
Duration of Mechanical ventilation | upto one month
  Total time of Mechanical ventilation required by the patient
Duration of PICU stay | upto one month
  Total Duration of stay in PICU
Duration of Hospital stay. | upto one month
  Total duration of Hospital stay in wards except PICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Mustahsin khalil Ahmad, MBBS, Principal Investigator — KEMU Lahore
Locations (1):
- King Edward Medical University Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNally JD, Menon K, Chakraborty P, Fisher L, Williams KA, Al-Dirbashi OY, Doherty DR; Canadian Critical Care Trials Group. The association of vitamin D status with pediatric critical illness. Pediatrics. 2012 Sep;130(3):429-36. doi: 10.1542/peds.2011-3059. Epub 2012 Aug 6. PMID 22869837
- [Background] McNally JD, Iliriani K, Pojsupap S, Sampson M, O'Hearn K, McIntyre L, Fergusson D, Menon K. Rapid normalization of vitamin D levels: a meta-analysis. Pediatrics. 2015 Jan;135(1):e152-66. doi: 10.1542/peds.2014-1703. Epub 2014 Dec 15. PMID 25511115
- [Background] Hossain N, Khanani R, Hussain-Kanani F, Shah T, Arif S, Pal L. High prevalence of vitamin D deficiency in Pakistani mothers and their newborns. Int J Gynaecol Obstet. 2011 Mar;112(3):229-33. doi: 10.1016/j.ijgo.2010.09.017. Epub 2011 Jan 17. PMID 21247568
- [Background] Mahmood K, Akhtar ST, Talib A, Haider I. Vitamin-D status in a population of healthy adults in Pakistan. Pak J Med Sci. 2009;25(4):545-50.
- [Background] Riaz H, Finlayson AE, Bashir S, Hussain S, Mahmood S, Malik F, Godman B. Prevalence of Vitamin D deficiency in Pakistan and implications for the future. Expert Rev Clin Pharmacol. 2016;9(2):329-38. doi: 10.1586/17512433.2016.1122519. Epub 2016 Jan 13. PMID 26582317
- [Background] Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Munch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial. JAMA. 2014 Oct 15;312(15):1520-30. doi: 10.1001/jama.2014.13204. PMID 25268295
- [Background] McNally D, Amrein K, O'Hearn K, Fergusson D, Geier P, Henderson M, Khamessan A, Lawson ML, McIntyre L, Redpath S, Weiler HA, Menon K; Canadian Critical Care Trials Group. Study protocol for a phase II dose evaluation randomized controlled trial of cholecalciferol in critically ill children with vitamin D deficiency (VITdAL-PICU study). Pilot Feasibility Stud. 2017 Dec 8;3:70. doi: 10.1186/s40814-017-0214-z. eCollection 2017. PMID 29234503
- [Background] Angurana SK. Serum Vitamin D Status and Outcome among Critically Ill Children Admitted to the Pediatric Intensive Care Unit in South India: Correspondence. Indian J Pediatr. 2016 Aug;83(8):910-1. doi: 10.1007/s12098-015-1992-z. Epub 2016 Jan 14. No abstract available. PMID 26762331
- [Background] Madden K, Feldman HA, Smith EM, Gordon CM, Keisling SM, Sullivan RM, Hollis BW, Agan AA, Randolph AG. Vitamin D deficiency in critically ill children. Pediatrics. 2012 Sep;130(3):421-8. doi: 10.1542/peds.2011-3328. Epub 2012 Aug 6. PMID 22869836
- [Background] Han JE, Jones JL, Tangpricha V, Brown MA, Brown LAS, Hao L, Hebbar G, Lee MJ, Liu S, Ziegler TR, Martin GS. High Dose Vitamin D Administration in Ventilated Intensive Care Unit Patients: A Pilot Double Blind Randomized Controlled Trial. J Clin Transl Endocrinol. 2016 Jun;4:59-65. doi: 10.1016/j.jcte.2016.04.004. Epub 2016 May 5. PMID 27419080
- [Background] Amrein K, Litonjua AA, Moromizato T, Quraishi SA, Gibbons FK, Pieber TR, Camargo CA Jr, Giovannucci E, Christopher KB. Increases in pre-hospitalization serum 25(OH)D concentrations are associated with improved 30-day mortality after hospital admission: A cohort study. Clin Nutr. 2016 Apr;35(2):514-521. doi: 10.1016/j.clnu.2015.03.020. Epub 2015 Apr 14. PMID 25935851
- [Background] Amrein K, Sourij H, Wagner G, Holl A, Pieber TR, Smolle KH, Stojakovic T, Schnedl C, Dobnig H. Short-term effects of high-dose oral vitamin D3 in critically ill vitamin D deficient patients: a randomized, double-blind, placebo-controlled pilot study. Crit Care. 2011;15(2):R104. doi: 10.1186/cc10120. Epub 2011 Mar 28. PMID 21443793
- [Background] Williams S, Heuberger R. Outcomes of Vitamin D Supplementation in Adults Who are Deficient and Critically Ill: A Review of the Literature. Am J Ther. 2016 Nov/Dec;23(6):e1890-e1902. doi: 10.1097/MJT.0000000000000281. PMID 26164022
- [Background] Gandhi J, Sangareddi S, Varadarajan P, Suresh S. Pediatric index of mortality 2 score as an outcome predictor in pediatric Intensive Care Unit in India. Indian J Crit Care Med. 2013 Sep;17(5):288-91. doi: 10.4103/0972-5229.120320. PMID 24339640
- [Background] Greenbaum LA. Rickets and Hypervitaminosis. In: Kliegman RM, Stanton BF, Geme III JW, Schor NF. (eds). Nelson Textbook Of Pediatrics. 20th ed. Philadelphia: Elsevier; 2016. p.331-38.
- [Background] Balasubramanian S, Dhanalakshmi K, Amperayani S. Vitamin D deficiency in childhood-a review of current guidelines on diagnosis and management. Indian Pediatr. 2013 Jul;50(7):669-75. doi: 10.1007/s13312-013-0200-3. PMID 23942432